CLINICAL TRIAL: NCT02805595
Title: A Single Center Clinical Trial to Evaluate the Effect of Sclerotherapy on Fistulas and Sinus Tracts in Adult Patients With Hidradenitis Suppurativa
Brief Title: Effect of Sclerotherapy on Fistulas and Sinus Tracts in Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Martina Porter, Instructor in Dermatology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001274
Record Dates: First submitted 2016-06-10; First posted 2016-06-20 (Estimated); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypertonic Saline (Experimental): 23.4% Hypertonic Saline injection(s) with a maximum of 0.4cc per treatment. If necessary every two weeks, with a maximum of three treatments.
  Interventions: Drug: 23.4% Hypertonic saline

INTERVENTIONS:
Drug: 23.4% Hypertonic saline — Saline Injections
  Other Names: 23.4% sodium chloride

SUMMARY:
This study evaluates the effect of hypertonic saline 23.4% injection in fistulas or sinus tracts in adult patients with hidradenitis suppurativa.

DETAILED DESCRIPTION:
The clinical effect of the hypertonic saline treatment will be evaluated with Physician Assessments at week 2 (t=2), week four (t=4) and week 8 (t=8) and compared with the first visit (baseline) (t=0). If necessary, subjects will be eligible to receive another hypertonic saline injected in week 2 and/or week 4, with a maximum of three injections. Simultaneously improvement will be assessed by ultrasound if possible, using the Philips Lumify Ultrasound Device, and by patients using HS Improvement Assessments. Pain and stinging during treatment sessions will be monitored using numeric rating scales (NRS). For monitoring quality of life the DLQI will be used.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects are at least 18 years of age or older
* A confirmed diagnosis of HS disease
* Presence of inflammatory HS lesion(s) and one or more fistula(s) or sinus tracts

Exclusion Criteria:

* Receiving any other kind of treatment for fistulas including introduction of anti-inflammatory systemic therapy such as prednisone or adalimumab within the prior month.
* Are participating in another study using an investigational agent or procedure during participation in this study.
* Are currently pregnant or planning to get pregnant during the study.
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martina Porter, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypertonic Saline
Started | 21
Completed | 17
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Demographic data was measured for all pariticipants, outcome measures were measured for only 17 completed subjects who had data for all visits. Physician assessment were only reported for 16sujbects
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.85 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: HS Physician Local Improvement Assessment - PAIN
Description: Percent change in clinical efficacy will be measured by Physician Assessments: HS Physician Local Improvement Assessment. Scale allows physician to score multiple HS symptoms on a scale from 'extremely worse' to 'very much improved'.
  Physicians rated characteristics associated with fistula severity as "improved", "no change", "worsened": overall clinical state of HS in treated area, pain, fluid leakage from fistula, erythema, tenderness on palpation, swelling, hardness of skin, hotness of skin, and odor.
Time Frame: Baseline and Visit 4 (week 8)
Population: 16 subjects completed the study and had percent score data for Baseline and Visit 4 comparison
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 16
Participants
  Improved | 7
  No Change | 7
  Worsened | 2

2. Primary Outcome: HS Physician Local Improvement Assessment - Fluid Leakage From Fistula
Description: as for outcome 1
Time Frame: Baseline and Visit 4 (week 8)
Population: 15subjects completed the study and had percent score data for Baseline and Visit 4 comparison. Not every subject had all fistula characteristic which is why total value is different for each separate characteristic.
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 15
Participants
  Improved | 9
  No Change | 5
  Worsened | 1

3. Primary Outcome: HS Physician Local Improvement Assessment - Erythema
Description: as for outcome 1
Time Frame: Baseline and Visit 4 (week 8)
Population: 16subjects completed the study and had percent score data for Baseline and Visit 4 comparison. Not every subject had all fistula characteristic which is why total value is different for each separate characteristic.
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 16
Participants
  Improved | 11
  No Change | 3
  Worsened | 2

4. Primary Outcome: HS Physician Local Improvement Assessment - Tenderness
Description: as for outcome 1
Time Frame: Baseline and Visit 4 (week 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 16
Participants
  Improved | 7
  No Change | 6
  Worsened | 3

5. Primary Outcome: HS Physician Local Improvement Assessment - Swelling
Description: as for outcome 1
Time Frame: Baseline and Visit 4 (week 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 16
Participants
  Improved | 10
  No Change | 5
  Worsened | 1

6. Primary Outcome: HS Physician Local Improvement Assessment - Hardness of Skin
Description: as for outcome 1
Time Frame: Baseline and Visit 4 (week 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 16
Participants
  Improved | 4
  No Change | 5
  Worsened | 7

7. Primary Outcome: HS Physician Local Improvement Assessment - Hotness of Skin
Description: as for outcome 1
Time Frame: Baseline and Visit 4 (week 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 16
Participants
  Improved | 3
  No Change | 12
  Worsened | 1

8. Primary Outcome: HS Physician Local Improvement Assessment - Odor
Description: as for outcome 1
Time Frame: Baseline and Visit 4 (week 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 16
Participants
  Improved | 5
  No Change | 10
  Worsened | 1

9. Secondary Outcome: Numeric Rating Scale for Stinging
Description: Self-reported median stinging intensity during and directly after treatment with Hypertonic saline injections.
  Pain with a score of 1 (no stinging at all) to 10 (worst possible stinging).
Time Frame: Baseline and visit 4 (week 8)
Population: Median score for Baseline and Visit 4 visits for 15 subjects who completed both visits.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 15
score on a scale
  Baseline | 5 (2.4)
  visit 4 | 5 (2.7)

10. Secondary Outcome: Numeric Rating Scale for Pain
Description: Self-reported median pain intensity during and directly after treatment with Hypertonic saline injections.
  Pain with a score of 1 (no pain at all) to 10 (worst possible pain).
Time Frame: Baseline and visit 4 (week 8)
Population: Baseline and Visit 4 pain scores were analyzed for 15 subjects who reported data for both visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 15
score on a scale
  Baseline | 3 (2.14)
  Visit 4 | 6 (2.54)

11. Secondary Outcome: Length of Fistula
Description: Measuring the length and the lumen of the fistulas using ultrasound if possible.
Time Frame: Baseline and visit 4 (week 8)
Population: Data was not analyzed or collected since measuring length of fistulas through ultrasound seemed not feasible. Measurement had to be taken from precise location at each visit for it to be accurate, but the fistula changed shape between visits which made is impossible to use these measures as an evaluation.
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 0

12. Secondary Outcome: Dermatology Life Quality Index
Description: Number of subjects improving based upon patient-reported outcomes The Dermatology Life Quality Index (DLQI) is a validated general dermatology questionnaire that consists of 10 items that assess subject health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment)
  The scoring of each question is as follows:
  Very much scored = 3 points, A lot scored = 2 points, A little scored = 1, Not at all scored = 0 points, Not relevant scored = 0 points, Question 7, 'prevented work or studying' scored = 3 points. The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 (meaning maximum impact on quality of life) and a minimum of 0 (meaning no impact of skin disease on quality of life). The higher the score, the more quality of life is impaired.
  0-1 = No effect on patient's life, 2-5 = Small effect, 6-10 = Moderate effect, 11-20 = Very large effect, 21-30 = Extremely large effect.
Time Frame: Baseline and visit 4 (week 8)
Population: DLQI score for subjects who had data for baseline and visit 4 (final visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 17
score on a scale
  Baseline | 9.14 (5.83)
  Visit 4 | 6.0 (5.62)

13. Secondary Outcome: HS Patient Local Improvement Assessment - Pain
Description: Percent change in Patient improvement assessment about state of the disease from baseline to visit 4. Scale allows physician to score multiple HS symptoms on a scale from 'extremely worse' to 'very much improved'.
  Patients rated characteristics associated with fistula severity as "improved", "no change", "worsened": Overall disease state of HS in treated area, pain, fluid leakage from fistula, erythema, tenderness on palpation, swelling, hardness of skin, hotness of skin, and odor.
Time Frame: Baseline to Visit 4 (week 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 16
Participants
  Improved | 13
  no change | 1
  worsened | 2

14. Secondary Outcome: HS Patient Local Improvement Assessment - Fluid From Fistula
Description: as for outcome 13
Time Frame: Baseline and Visit 4 (week 8)
Population: 17subjects completed the study and had percent score data for Baseline and Visit 4 comparison. Not every subject had all fistula characteristic which is why total value is different for each separate characteristic.
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 17
Participants
  Improved | 14
  No Change | 0
  Worsened | 3

15. Secondary Outcome: HS Patient Local Improvement Assessment - Erythema
Description: as for outcome 13
Time Frame: Baseline and Visit 4 (week 8)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 17
Participants
  Improved | 13
  No Change | 2
  Worsened | 2

16. Secondary Outcome: HS Patient Local Improvement Assessment - Tenderness
Description: as for outcome 13
Time Frame: Baseline and Visit 4 (week 8)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 17
Participants
  Improved | 15
  No Change | 1
  Worsened | 1

17. Secondary Outcome: HS Patient Local Improvement Assessment - Swelling
Description: as for outcome 13
Time Frame: Baseline and Visit 4 (week 8)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 17
Participants
  Improved | 15
  No Change | 2
  Worsened | 0

18. Secondary Outcome: HS Patient Local Improvement Assessment - Hardness of Skin
Description: as for outcome 13
Time Frame: Baseline and Visit 4 (week 8)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 17
Participants
  Improved | 10
  No Change | 3
  Worsened | 4

19. Secondary Outcome: HS Patient Local Improvement Assessment - Hotness of Skin
Description: as for outcome 13
Time Frame: Baseline and Visit 4 (week 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 16
Participants
  Improved | 8
  No Change | 8
  Worsened | 0

20. Secondary Outcome: HS Patient Local Improvement Assessment - Odor
Description: as for outcome 13
Time Frame: Baseline and Visit 4 (week 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertonic Saline
Number analyzed (Participants) | 16
Participants
  Improved | 10
  No Change | 3
  Worsened | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 8 weeks for each subject.
Description: Definition doe snot differ, expected adverse events listed in the ICF were not collected or reported as per institution IRB guidelines
Arm/Group | Hypertonic Saline
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
Study limitations include 1) small sample size and lack of a control group. 2) the lack of an established scoring system for assessing improvement in individual fistulas. 3) We were unable to determine full fistula dimensions over time with ultrasound. 4) This was a single team of clinical investigators; therefore, treatment efficacy cannot be assessed between study investigators who were not trained by the original investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT02805595/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT02805595/ICF_001.pdf